CLINICAL TRIAL: NCT04251000
Title: Joovv for Seasonal Affective Disorder
Brief Title: Infrared Photomodulation Therapy for Seasonal Affective Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProofPilot (Industry)
Collaborators: Joovv (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2393
Record Dates: First submitted 2020-01-25; First posted 2020-01-31 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-01

CONDITIONS: Seasonal Affective Disorder
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Intervention Model Description: Single arm pilot study
Masking Description: This is a single arm unblineded effort.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Joovv Pilot Experimenta Arm (Experimental): Individuals will receive 90 day access to the Joovv infrared mini light device.
  Interventions: Device: Joovv Mini

INTERVENTIONS:
Device: Joovv Mini — the smallest photomodulation device in the Joovv infrared light product line.

SUMMARY:
During winter months in northern latitudes use of Joovv device on self-reported non-clinical mental health (aka mood), sleep and energy levels. Participants will also submit Withings and Oura activity and sleep data.

ELIGIBILITY:
Inclusion Criteria:

* history of mental health issues including clinical depression
* US based
* reasonably active individuals (self report run/gym 3x per week or more)

Exclusion Criteria:

* average daily high temperature in zipcode above 60 degrees through end of March

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
change self report mood as assessed by Warwick Edinburgh sleep scale | Baseline to 90 day
  non clinical measures of mood controlled for environmental temperature and daylight
Change in Sleep Duration and Sleep Quality as measured by consumer connected health device | Baseline to 90 day
  Measures of sleep and sleep quality as by a Withings or Oura Ring connected health device
Change in activity levels as measured by consumer connected health devices | Baseline to 90 day
  Measures of activity levels as by WIthings our Oura connected health devices

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Virtual Study: https://proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
currently no plans.